CLINICAL TRIAL: NCT02281747
Title: Frequency and Complications of Major Orthopedic Procedures in Medicare Beneficiaries and Other Databases
Brief Title: Frequency and Complications of Major Orthopedic Procedures in Medicare Beneficiaries
Status: Active, not recruiting | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999915010; 15-AR-N010
Record Dates: First submitted 2014-10-31; First posted 2014-11-04 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-12-19

CONDITIONS: Rheumatoid Arthritis; Ankylosing Spondylitis
Keywords: Biologic Therapy; Rheumatoid Arthritis; Arthroplasty; Natural History
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- affected with arthritis: arthritis may be either rheumatoid, osteoarthritis, or ankylosing spondylitis
- unaffected with arthritis: in some analyses, the comparison is by arthritis status. in other analyses, it is within arthritis status by clinically relevant subgroups.

SUMMARY:
Background:

- Orthopedic procedures are common in the United States. These include joint replacement and spine surgeries. Researchers want to study data about these procedures over time. They want to see if treatment has gotten better. They also want to find ways to change the care that people get before and after they have these procedures. These changes may lower the risk of problems people can have during and after treatment. They may also improve people s results.

Objectives:

- To study a series of questions about surgery, medicine, treatments, and outcomes for orthopedic procedures.

Eligibility:

- Data from the U.S. Centers for Medicare and Medicaid Services from 1999 to 2015.

Design:

* Researchers will look at data for people ages 20-100.
* No new participants will be used in this study.
* The study will last 6 years.

DETAILED DESCRIPTION:
Major orthopedic procedures, including total joint replacement and spine surgeries, are among the most common procedures in the population. Learning about how often these surgeries are performed can give indications of whether the treatment of arthritis and other musculoskeletal conditions has been improving over time. Learning about the complications associated with these surgeries can give indications about ways to alter the care of patients before and after surgeries that may decrease the risk of complications and improve patient outcomes. We will analyze Medicare and Medicaid data from 1999 to 2015 to examine a series of questions, including whether the use of joint replacement surgery has changed over time among patients with rheumatoid arthritis and ankylosing spondylitis, to see if rheumatoid arthritis medications are associated with some types of surgical complications, to see if anticoagulation medication after joint replacement is associated with the risk of complications, to see if regional differences in surgery rates can be explained by differences in patient characteristics, and to determine the surgical treatment for hip fractures that is associated with the fewest long-term complications. From the Framingham Heart Study Cohort, we will study the changes in the incidence of hip fractures and the risk factors for osteoporosis over time.

ELIGIBILITY:
* Subjects will be either Medicare or Medicaid beneficiaries with available claims from 1999 to 2015. For projects requiring detailed medication information, inclusion will be limited to those with Part D claims from 2006 to 2015. Eligibility for each project will be based on claims for the appropriate disease (e.g. RA) or procedure (e.g. hip arthroplasty).

Medicare beneficiaries will be excluded (or censored) if they do not have both Part A and Part B coverage, or enrolled in Medicare Advantage plans (Part C), as detailed claims for these beneficiaries are not available. We will also exclude dual-eligible (Medicare and Medicaid recipients) as these subjects have distinct clinical conditions (e.g. blindness) that distinguishes them from most Medicare beneficiaries. There will be no exclusions based on gender, race, ethnicity, or cognitive impairment.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medicare (1999 to 2015) and Medicaid (1999 to 2015) beneficiaries
Sampling Method: Non-Probability Sample
Enrollment: 521292 (Actual)
Dates: Start 2014-10-24 (Actual); Primary Completion 2029-05-30 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Complications | 30 days
  Complications

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Colbert, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS), 9, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
undecided yet